CLINICAL TRIAL: NCT03729076
Title: Crystalloid Versus Colloid Rapid Co-load in Parturients Receiving Prophylactic Phenylephrine Infusion During Cesarean Delivery Under Spinal Anesthesia
Brief Title: Crystalloid Versus Colloid Rapid Co-load for Cesarean Delivery Under Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-1807-152-961
Record Dates: First submitted 2018-10-28; First posted 2018-11-02 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Pregnancy; Cesarean Delivery; Hypotension
MeSH Terms: conditions — Hypotension | interventions — Crystalloid Solutions; Colloids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crystalloid (Experimental): Patients will receive rapid co-load of plasma solution A (PSA) 10ml/kg, from the initiation of spinal anesthesia.
  Interventions: Other: Crystalloid
- Colloid (Active Comparator): Patients will receive rapid co-load of 6% volulyte (HES in acetated electrolyte) 10ml/kg, from the initiation of spinal anesthesia.
  Interventions: Other: Colloid

INTERVENTIONS:
Other: Crystalloid — Patients will receive the rapid co-loading with plasma solution A (PSA) 10ml/kg, from the initiation of spinal anesthesia, within 10 minutes.
  Arms: Crystalloid
Other: Colloid — Patients will receive the rapid co-loading with 6% volulyte (HES in acetated electrolyte) 10ml/kg, from the initiation of spinal anesthesia, within 10 minutes.
  Arms: Colloid

SUMMARY:
The study aims to compare crystalloid co-loading and colloid co-loading in parturients receiving prophylactic phenylephrine infusion during cesarean delivery in terms of the incidence of hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, full-term parturients who scheduled to undergo elective cesarean delivery under spinal anesthesia.

Exclusion Criteria:

* multiple pregnancy

  * gestational age < 36 weeks

    * preexisting or pregnancy-induced hypertension

      * Morbid cardiovascular impairments

        * Cerebrovascular disease

          ⑥ Known fetal anomaly

          ⑦ Contraindications to spinal anesthesia

          ⑧ Any sign of onset of labor

          ⑨ Body weight < 45 kg or body weight > 90 kg

          ⑩ Height < 145cm or height > 180cm

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Parturients
Enrollment: 100 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-12 (Actual)

PRIMARY OUTCOMES:
Incidence of maternal hypotension | during the time period from induction of spinal anesthesia until delivery
  defined as: Systolic Blood Pressure (SBP) < 80% of baseline SBP

SECONDARY OUTCOMES:
incidence of severe hypotension | during the time period from induction of spinal anesthesia until delivery
  defined as: Systolic Blood Pressure (SBP) < 70% of baseline SBP
incidence of symptomatic hypotension | during the time period from induction of spinal anesthesia until delivery
  defined as: hypotension plus nausea and/or vomiting and/or dizziness and/or breathlessness
incidence of bradycardia | during the time period from induction of spinal anesthesia until delivery
  Heart Rate (HR) <50 bpm
incidence of Hypertension | during the time period from induction of spinal anesthesia until delivery
  Systolic Blood Pressure (SBP)> 120% of baseline SBP
Minimum recorded Systolic Blood Pressure (Minimum SBP) | during the time period from induction of spinal anesthesia until delivery
  The lowest recorded SBP during the time period from induction of spinal anesthesia until delivery
Minimum recorded Heart Rate (Minimum HR) | during the time period from induction of spinal anesthesia until delivery
  The lowest recorded HR during the time period from induction of spinal anesthesia until delivery
Cumulative duration of hypotension | during the time period from induction of spinal anesthesia until delivery
  duration of hypotension, minutes
Onset time of hypotension | during the time period from induction of spinal anesthesia until delivery
  Time from the induction of spinal anesthesia until the first event of hypotension occur
Total phenylephrine use | during the time period from induction of spinal anesthesia until delivery
  Cumulative dose of phenylephrine administered via continuous infusion, mcg
Rescue phenylephrine use | during the time period from induction of spinal anesthesia until delivery
  number of patients who require the rescue use of phenylephrine
Rescue ephedrine use | during the time period from induction of spinal anesthesia until delivery
  number of patients who require the rescue use of ephedrine
Atropine use | during the time period from induction of spinal anesthesia until delivery
  number of patients who require the rescue use of atropine
Incidence of nausea, vomiting | during the time period from induction of spinal anesthesia until delivery
  The incidence of nausea, vomiting
Incidence of dizziness, breathlessness | during the time period from induction of spinal anesthesia until delivery
  The incidence of dizziness, breathlessness
Cutaneous stellate ganglion sympathetic activity | during the time period from induction of spinal anesthesia until delivery
  noninvasive recording of skin sympathetic nerve activity (SKNA) using conventional ECG electrodes
Apgar Score, 1 min, 5 min (fetal outcome) | 1 min, 5 min after delivery
  Apgar Score of delivered baby. The Apgar score is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. The five criteria are the Appearance, Pulse, Grimace, Activity, and Respiration. Each is scored on a scale of 0 to 2, with 2 being the best score. The test is done at 1 and 5 minutes after birth.
Umbilical arterial pH | immediately after delivery
  pH of Umbilical Arterial blood gas analysis (ABGA) (fetal outcome)
Umbilical arterial base excess | immediately after delivery
  base excess of Umbilical ABGA (fetal outcome), mmol/L
Umbilical arterial partial oxygen pressure (PO2) | immediately after delivery
  partial oxygen pressure of Umbilical ABGA (fetal outcome), mmHg
Umbilical arterial carbon dioxide partial pressure (PCO2) | immediately after delivery
  carbon dioxide partial pressure of Umbilical ABGA (fetal outcome), mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD, PhD, Principal Investigator — Seoul National University Hospital, Seoul National University College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kinsella SM, Carvalho B, Dyer RA, Fernando R, McDonnell N, Mercier FJ, Palanisamy A, Sia ATH, Van de Velde M, Vercueil A; Consensus Statement Collaborators. International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia. Anaesthesia. 2018 Jan;73(1):71-92. doi: 10.1111/anae.14080. Epub 2017 Nov 1. No abstract available. PMID 29090733
- [Background] Ripolles Melchor J, Espinosa A, Martinez Hurtado E, Casans Frances R, Navarro Perez R, Abad Gurumeta A, Calvo Vecino JM. Colloids versus crystalloids in the prevention of hypotension induced by spinal anesthesia in elective cesarean section. A systematic review and meta-analysis. Minerva Anestesiol. 2015 Sep;81(9):1019-30. Epub 2014 Dec 11. PMID 25501602
- [Background] Tawfik MM, Tarbay AI, Elaidy AM, Awad KA, Ezz HM, Tolba MA. Combined Colloid Preload and Crystalloid Coload Versus Crystalloid Coload During Spinal Anesthesia for Cesarean Delivery: A Randomized Controlled Trial. Anesth Analg. 2019 Feb;128(2):304-312. doi: 10.1213/ANE.0000000000003306. PMID 29461392
- [Background] Doytchinova A, Hassel JL, Yuan Y, Lin H, Yin D, Adams D, Straka S, Wright K, Smith K, Wagner D, Shen C, Salanova V, Meshberger C, Chen LS, Kincaid JC, Coffey AC, Wu G, Li Y, Kovacs RJ, Everett TH 4th, Victor R, Cha YM, Lin SF, Chen PS. Simultaneous noninvasive recording of skin sympathetic nerve activity and electrocardiogram. Heart Rhythm. 2017 Jan;14(1):25-33. doi: 10.1016/j.hrthm.2016.09.019. Epub 2016 Sep 23. PMID 27670627